CLINICAL TRIAL: NCT00449995
Title: Confocal Laserscanning Microscopy for Detection of Barretts Esophagus. A Blinded Multi-Center Study.
Brief Title: Confocal Laserscanning Microscopy for Detection of Barretts Esophagus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Charite University, Berlin, Germany (Other); Technische Universität Dresden (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1129/04
Record Dates: First submitted 2007-02-23; First posted 2007-03-21 (Estimated); Last update posted 2008-12-24 (Estimated); Status verified 2008-12

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus | interventions — Microscopy, Confocal

INTERVENTIONS:
Procedure: confocal laser microscopy

SUMMARY:
Four quadrant biopsies in regular ranges is the goldstandard in monitoring this disease. The ideal situation for the endoscopist is to visualize cellular structures, which implies having microscopic imaging available. A potential candidate to fill this gap could be confocal fluorescence microscopy (Cellvizio®-GI and Mauna Kea Technologies). To compare the gold standard with the confocal fluorescence microscopy for detection of metaplastic - or intraepithelial neoplastic changes of barrett-suspicious esophageal mucosa this study has been initiated.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 80 years
* regular esophagogastroduodenoscopy for patients with known barrett esophagus (at least stadium C0M1)
* patients presenting for endoscopic mucosectomy with intraepithelial neoplastic changes <1cm
* patients presenting with suspected intraepithelial neoplastic changes
* patients receiving acid suppressive therapy in standard dose for at least 4 weeks

Exclusion Criteria:

* no informed consent
* thrombocytopenia, quick <50%, PTT >50 sec
* patients with coronary heart disease or existent valve plasties
* women with potential pregnancy
* patients with chronic renal failure
* patients with allergies
* patients with chronic obstructive pulmonary disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-07 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
diagnostic accuracy of confocal laser scanning microscopy for detection of metaplasia or neoplasia in Barrett´s esophagus

SECONDARY OUTCOMES:
inter- and intra observer variability for confocal laser scanning microscopy

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Meining, MD, Principal Investigator — Technical University Munich
Locations (1):
- 2nd department of the Medical Clinic of the Technical University Munich, Munich, Bavaria, Germany